CLINICAL TRIAL: NCT02608944
Title: Comparison of New MRI Methods for Quantitative Assessment of Myocardial Perfusion With Quantitative PET Perfusion Imaging
Brief Title: Comparison of Quantitative MRI Perfusion Methods With Quantitative PET Perfusion Imaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: MRI perfusion techniques development took longer than expected.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Edward DiBella, Ph.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB 58133
Record Dates: First submitted 2015-11-10; First posted 2015-11-20 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: MRI Scans
MeSH Terms: interventions — Adenosine; regadenoson; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI perfusion vs. PET Imaging perfusion (Experimental): Adenosine Regadenoson O-15 labeled radioactive water MRI PET Imaging
  Interventions: Drug: Adenosine; Drug: Regadenoson; Drug: O-15 labeled radioactive water; Device: MRI; Device: PET Imaging

INTERVENTIONS:
Drug: Adenosine — Adenosine: 0.14mg/kg/min for 6 min. IV injection for MRI perfusion
  Other Names: Adenoscan; Adenocard
Drug: Regadenoson — Regadenoson: 0.4mg in 5ml, given as a rapid (10 seconds) IV injection for MRI perfusion.
  Other Names: Lexiscan
Drug: O-15 labeled radioactive water — O-15 labeled radioactive water: Up to 50mCi IV injection at rest and again at hyperemia for PET Imaging
  Other Names: O-15 water
Device: MRI — Pass dynamic contrast enhanced MRI scans will be performed at rest and during hyperemia caused by either adenosine infusion or regadenoson
Device: PET Imaging — Quantitative PET imaging with O-15 labeled radioactive water will be given at a different day.
  Other Names: Positron Emission Tomography Imaging

SUMMARY:
This work seeks to develop, evaluate and use new MRI methods for non-invasive quantitative assessment of myocardial perfusion and perfusion reserve (MPR), and to compare with quantitative PET imaging.

DETAILED DESCRIPTION:
This project aims to determine the validity of quantitative MRI perfusion methods by comparison with quantitative PET imaging. First pass dynamic contrast enhanced MRI scans will be performed at rest and during hyperemia caused by either adenosine infusion or regadenoson. After custom reconstruction and post-processing the data will be fit to a compartment model and quantitative perfusion and MPR values obtained.

On another day, the subjects will have quantitative PET imaging with O-15 labeled radioactive water. This will be done at rest and hyperemia caused by either adenosine or regadenoson. A low dose CT scan will be acquired to perform attenuation correction of the PET images. The images will be reconstructed and processed as reported in the literature to provide reference standard perfusion and MPR values. These values will be compared with those obtained by MRI.

ELIGIBILITY:
* Inclusion Criteria:

  * All participants will be over the age of 18 and able to provide consent
  * Both healthy and subjects with cardiac disease (including atrial fibrillation but not required) will be recruited.
* Exclusion Criteria:

  * Critically ill patients, patients on ventilators, patients with unstable angina or with hypotension, asthmatics, and other patients whose medical care or safety may be at risk from undergoing an MRI examination will be excluded.
  * Patients with claustrophobia will also be excluded from the study if this cannot be controlled with standard methods (valium or benadryl).
  * Patients with contraindication to MRI (pacemaker, metal implants, or certain types of heart valves),
  * pregnant patients, minors, mentally disabled patients and prisoners will be excluded from this study. (All criteria apply to patients and normal volunteers).
  * Gadolinium nephrotoxicity will be addressed by having patients with abnormal kidney function (GFR<30) excluded from the study due to the (very small) risk associated with gadolinium contrast agents. This threshold may be modified, depending on practices determined by the Radiology Department and the IRB.
  * Patients with a known allergy or contraindication to Adenosine and/or Regadenoson will be excluded from stress (hyperemia) cohorts.
  * All participants that will receive a stress agent will refrain from consuming caffeine for at least 12 hours prior to each study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09-30 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion values from MRI | The scan will take ~1-2 hours. The MRI will be done within 2 months of the PET scan.
  Myocardial perfusion in segments and coronary territories will be computed in ml/min/g from the dynamic MRI data. The perfusion values will be compared to PET data to determine how similar the values are.
Myocardial perfusion values from PET | The scan will take ~1-2 hours. The PET scan will be done within 2 months of the MRI.
  Myocardial perfusion in segments and coronary territories will be computed in ml/min/g from the dynamic PET data. The perfusion values will be compared to MRI data to determine how similar the values are.

CONTACTS AND LOCATIONS:
Overall Officials: Edward DiBella, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Radiology Research, Salt Lake City, Utah, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT02608944/Prot_SAP_000.pdf